CLINICAL TRIAL: NCT05350371
Title: Evaluation of Pirfenidone as a Therapy in Patients With Predicted Moderate to Severe Acute Pancreatitis
Brief Title: Safety and Tolerability of Pirfenidone in Acute Pancreatitis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Nikhil Bush Jayaram, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-300008875
Record Dates: First submitted 2022-03-23; First posted 2022-04-28 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-06

CONDITIONS: Pancreatitis, Acute
MeSH Terms: conditions — Pancreatitis | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Experimental)
  Interventions: Drug: Placebo
- Pirfenidone Treatment (Experimental)
  Interventions: Drug: Pirfenidone Oral Tablet

INTERVENTIONS:
Drug: Pirfenidone Oral Tablet — Patients in the pirfenidone treatment arm will be given pirfenidone 267mg tablet, tid for 1 day followed by dose escalation to two 267 mg tablet tid for 6 days. Thus, the treatment will be for total of 7 days or till patients develop an adverse event that requires their participation in the study to be stopped.
  Arms: Pirfenidone Treatment
Drug: Placebo — The placebo tablets will be an exact replica of the pirfenidone tablet.
  Arms: Placebo

SUMMARY:
The goal of the current pilot clinical trial is to evaluate the safety and tolerability of pirfenidone in patients with predicted moderately severe and severe acute pancreatitis. Pirfenidone is currently approved by FDA for the treatment of idiopathic pulmonary fibrosis. Now, over 5 years of data has accumulated demonstrating safety of its use in humans. The investigators' preclinical data suggest that pirfenidone is very effective in reducing the severity of acute pancreatitis in animal models. Following are the objectives of the proposed clinical trial:

Primary Objective:

* To evaluate the safety and tolerability of pirfenidone, compared to placebo, in patients predicted to have moderately severe or severe AP.
* To evaluate the efficacy of pirfenidone in reducing the laboratory markers of inflammation and improving patient reported outcome measures.

Secondary Objective:

- To evaluate the efficacy of pirfenidone in reducing the severity of acute pancreatitis, as measured by well-defined endpoints.

DETAILED DESCRIPTION:
The study is a Randomized Pilot clinical trial evaluating safety and tolerability of pirfenidone in patients with predicted moderately severe to severe acute pancreatitis. There are built in secondary end-points for efficacy. The patients with acute pancreatitis, who present within 48h of establishment of the diagnosis, will be screened for exclusion and inclusion criteria and consented for the clinical trial. Patients with be randomized into placebo or pirfenidone arm and followed daily in-person, while in hospital, and by telephone once discharged from the hospital (weekly for 4 weeks, then monthly for up to 6 months) for study end points.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 - 85 years of age
2. Admitted to hospital for AP, defined by at least 2 of the following 3:

   1. amylase or lipase values, or both, that are greater than 3 times the upper limit of normal values
   2. characteristic cross-sectional imaging
   3. typical upper abdominal pain- acute onset of a persistent, severe, epigastric pain often radiating to the back
3. Patients identified, approached, and consented to administer study medication or placebo within 48 hours of diagnosis of AP.
4. Predicted to have MSAP or SAP by presence of one or more of the following criteria

   1. APACHE II ≥ 8
   2. Modified Glasgow or Imrie score ≥ 3
   3. CRP > 150 mg/dL
   4. PASS score > 140 at or within 48 hrs. of admission
   5. CT or MRI imaging suggesting pancreatic and/or peri-pancreatic necrosis

Exclusion Criteria:

1. Age < 18 or > 85 years
2. Body weight > 200 kg
3. Presentation to the medical attention > 48 h after diagnosis of AP
4. Inability to recruit, randomize and start the allocated treatment within 48h of start of pain
5. Ongoing AP or diagnosis of AP in previous 30 days
6. Chronic pancreatitis
7. Known hypersensitivity to pirfenidone
8. AST/ALT ≥ 2 times the upper normal limit.
9. Alkaline phosphatase ≥ 2 times the upper normal limit
10. Bilirubin higher than upper normal limit
11. Moderate to severe heart failure and/or coronary heart disease (New York Heart Association (NYHA) Functional Class III/IV)
12. On home oxygen or home mechanical ventilation
13. Advanced liver disease
14. Paralytic ileus or significant nausea and vomiting
15. Chronic Diarrhea
16. Immunosuppressive disorder or on immunosuppressive medications
17. Active or advanced malignancy
18. Known cancer that is end-stage with ongoing palliative care or for which palliative care is appropriate
19. Known established infection prior to the onset of acute pancreatitis
20. Known history of infective hepatitis
21. Known live vaccines or therapeutic infectious agents within one month of admission
22. Known pregnancy or lactation at the time of admission
23. Ongoing photosensitivity and rash
24. Women of childbearing potential who are not on oral or injectable contraceptives or IUDs and do not consent to practice abstinence for period of 4 weeks.
25. Known to be currently participating in a trial testing any investigational medicinal product or participation in a clinical study involving a medicinal product in the last three months
26. Alcohol or substance abuse in the past 2 years
27. Family or personal history of long QT syndrome ( > 500 msec)
28. Medications like fluvoxamine or sildanefil
29. Significant photosensitivity or new rash
30. Renal disease with GFR < 30
31. Any condition other than above that, in the opinion of the investigator, is likely to result in the death of the patient within the next 2 years
32. Any condition that, in the opinion of the investigator, might be significantly exacerbated by the known side effects associated with the administration of pirfenidone

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Development of anticipated or un-anticipated serious adverse events (class 3 or 4) | 6 months
  Development of anticipated or un-anticipated serious adverse events (class 3 or 4)
percentage of patients starting and completion of the planned drug treatment | 7 days
  percentage of patients starting and completion of the planned drug treatment
Changes in C-reactive protein (CRP), TNF-α, interleukin (IL)-6, IL-8 and IL-10 levels | 7 days
  Compared to base line
percentage of patients having decrease in PAN-PROMISE score by at least 10 points at 72h after initiation of the drug | 3 days
  Measurement of PAN-PROMISE score

SECONDARY OUTCOMES:
cumulative PAN-PROMISE score | 7
  total of the PAN-PROMISE over 7 days
cumulative PASS score | duration of admission
  total of PASS score during admission
PASS score at the time of discharge | duration of admission
  PASS score measurement
Composition outcome | 6 months
  total of development of new or worsening pancreatic or peri-pancreatic necrosis, death or major infection
Readmission and/or ER visits | within 30 days and within 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UAB, Birmingham, Alabama
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palathingal Bava E, George J, Tarique M, Iyer S, Sahay P, Gomez Aguilar B, Edwards DB, Giri B, Sethi V, Jain T, Sharma P, Vaish U, C Jacob HK, Ferrantella A, Maynard CL, Saluja AK, Dawra RK, Dudeja V. Pirfenidone increases IL-10 and improves acute pancreatitis in multiple clinically relevant murine models. JCI Insight. 2022 Jan 25;7(2):e141108. doi: 10.1172/jci.insight.141108. PMID 34847076
- [Derived] Bava EP, Jain T, Al-Obaidi M, Evans Z, Doto D, Vege SS, Dudeja V. Safety, tolerability and therapeutic efficacy of anti-inflammatory drug pirfenidone in acute pancreatitis patients: Protocol for a randomized pilot clinical trial. Pancreatology. 2025 Mar;25(2):214-220. doi: 10.1016/j.pan.2025.01.004. Epub 2025 Jan 13. PMID 39864969